CLINICAL TRIAL: NCT03972696
Title: OPTimizing Irradiation Through Molecular Assesment of Lymph Node After Primary Systemic Treatment
Acronym: OPTIMALIIa
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The inclusion rate of patients is too slow, so it is not possible to reach the estimated N.
Sponsor: Grupo de Investigación Clínica en Oncología Radioterapia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIC-RAD-2016-01
Record Dates: First submitted 2019-05-31; First posted 2019-06-04 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BA3S (Active Comparator): Radiotherapy (RT) will be administered, in the breast or thoracic wall, axillary levels I, II and III, and supraclavicular node areas, with optimization of the technique Intentional irradiation of lymph nodes: Patients will receive a total dose of 50 Gy in the whole breast and nodal areas (axillary I, II, III, and supraclavicular) with optimization of the technique, in daily fractions of 2 Gy and 5 fractions/week during 5 weeks.
  Interventions: Radiation: Irradiation
- BA2 (Experimental): RT will be administered, in the breast or thoracic wall and axillary levels I and II, with optimization of the technique Incidental irradiation of lymph nodes: Patients will receive a total dose of 50 Gy in the whole breast, but not aimed at nodal areas, with optimization of the technique, in daily fractions of 2 Gy and 5 fractions/week during 5 weeks.
  Interventions: Radiation: Irradiation

INTERVENTIONS:
Radiation: Irradiation — BA3S versus BA2 irradiation of lymphatic node areas, administered using a lineal accelerator, after 3D delimitation of the supraclavicular and axillary levels I, II and III. In both treatment arms, further tumoral bed boost will be allowed according to the investigator criteria, whether dose contribution to the nodal areas can be calculated. Due to its nature, interventions cannot be asked.

SUMMARY:
Breast cancer management integrating surgery, systemic therapy and radiation therapy tends to systemic treatment as the first therapeutic option, continuing afterwards by surgery and radiation therapy with the scope of decreasing the locoregional treatment. This strategy implies doubts about what should be the locoregional treatment, because many patients have remissions and a significant number of them a complete response. The responses are associated with better clinical outcome although there are doubts about they are a surrogate marker of survival.

Nodal irradiation after systemic treatment in patients with breast cancer it is under discussion, particularly in the case of patients with initial clinical involvement experiencing complete remission. For this reason, some groups decide irradiation of all nodal regions and others choose no irradiation of the lymph nodes at all. To clarify this discussion the present study is proposed.

The "One Step Nucleic Amplification" (OSNA) is a technique developed by Sysmex Corporation that allows a complete analysis of sentinel nodes and provides a quantification of the tumor marker Cytokeratin 19 (CK19) messenger ribonucleic acid (mRNA) in the sentinel node. The result is expressed by the Tumour Load as number of copies per microliter. This technique has shown its diagnostic ability both without primary systemic treatment and after primary systemic treatment, being more reproducible than conventional processes.

In spite of this, fits to mention that the studies of validation used to obtain the European Conformity (CE) mark only included patients without previous systemic treatment to the surgery.

DETAILED DESCRIPTION:
Breast cancer management integrating surgery, systemic therapy and radiation therapy tends to systemic treatment as the first therapeutic option, continuing afterwards by surgery and radiation therapy with the scope of decreasing the locoregional treatment. This strategy implies doubts about what should be the locoregional treatment, because many patients have remissions and a significant number of them a complete response. The responses are associated with better clinical outcome although there are doubts about they are a surrogate marker of survival.

According to a previous publication, in which the predictors of locoregional recurrence National Surgical Adjuvant Breast and Bowel Project 18 (NSABP18) and National Surgical Adjuvant Breast and Bowel Project 27 (NSABP27) studies are evaluated, both studies designed for viewing the value of neoadjuvant chemotherapy, good results of locoregional control are described, although in many cases radiotherapy was omitted or lymph node were not irradiated.

Therefore the need to nodal irradiation begins to be questioned, especially when they are negative after primary systemic treatment, regardless of their previous state. However the clinical guidelines recommend radiotherapy planning according to the previous stage. The problem is the local treatment indication is established based on the indications of irradiation without primary systemic therapy, as showed in retrospective studies, without the existence of randomized studies designed to analyze the role of radiotherapy in these circumstances. In the last American Society of Clinical Oncology (ASCO) preliminary results of a meta-analysis including three large studies of primary systemic treatment were presented.

Results show that irradiation improves local control in N1 patients achieving a complete remission, radiotherapy being an independent prognostic factor, in terms of locoregional control; however, they conclude that the optimal selection of patients remains unclear. The controversy remains, because there is no evidence to treat nodes after primary systemic therapy, whether there is a complete remission as if it does not, nor is it known that subgroup of patients may benefit more from local treatments. Long-term studies are needed to analyze this issue, leaving the decision being especially complicated in cases of clinically positive nodes experiencing a complete remission. The problem remains that often is not known exactly has been irradiated since, in many studies, irradiation is indicated at the discretion of the researcher.

Given these doubts, European Society conducted a survey to find out what was the attitude about these patients, and the findings shows that 75% of the centers irradiate in the N1 case. The American Society obtained similar results and in Spain 64% of respondents irradiate the lymph nodes. These three publications conclude that studies are needed to determine the importance of irradiation after primary systemic treatment and while waiting for these results, a consensus muts be reached as stated in ASCO 2015 summary.

The "One Step Nucleic Amplification" (OSNA) is a technique developed by Sysmex Corporation that allows a complete analysis of sentinel nodes and provides a quantification of the tumor marker CK19 mRNA in the sentinel node. The result is expressed by the Tumour Load as number of copies per microliter. This technique has shown its diagnostic ability both without primary systemic treatment and after primary systemic treatment, being more reproducible than conventional processes.

In spite of this, fits to mention that the studies of validation used to obtain the CE mark only included patients without previous systemic treatment to the surgery.

In summary, nodal irradiation after systemic treatment in patients with breast cancer it is under discussion, particularly in the case of patients with initial clinical involvement experiencing complete remission. For this reason, some groups decide irradiation of all nodal regions and others choose no irradiation of the lymph nodes at all. To clarify this discussion the present study is proposed.

ELIGIBILITY:
Inclusion Criteria:

* Infiltrating carcinoma of the breast.
* Metastatic lymph nodes (N1) at diagnosis, as determined histologically by Fine Needle Aspiration or Core Needle Biopsy.
* Primary systemic therapy (including antiestrogen or chemotherapy, and targeted therapies).
* Tumour surgery: tumorectomy, quadrantectomy or mastectomy.
* OSNA (ND) or - lymph nodes after primary systemic therapy.
* Age ≥ 18 years old.
* Karnofsky Index ≥ 70 %.
* Signed Informed Consent.

Exclusion Criteria:

* Lymphadenectomy.
* Bilateral breast cancer.
* Males.
* Previous thoracic irradiation therapy.
* Contraindications of radiotherapy (pregnancy, severe collagen diseases).
* Other neoplasms.
* Severe associated comorbidities that, according to the investigator criteria, may interfere with the study evaluations.
* Lymp nodes OSNA -(L), +, ++ after primary systemic therapy.
* Sentinel lymph node biopsy previous to the primary systemic therapy.
* Mammary internal chain affected.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
To show the non-inferiority of (BA2) compared to (BA3S), in terms of 5-years diseasefree survival (DFS), including the local, regional and distant disease free survival and excluding second neoplasms | 5 years
  The primary outcome will be the 5-years DFS. DFS is defined as the time from randomization to any breast cancer-related event, including local, regional or distant recurrence, or death from breast cancer.

SECONDARY OUTCOMES:
To compare the 5-years incidence of loco-regional tumor recurrence between BA2 and BA3S. | 5 Years
  Loco-regional recurrence during the 5-years follow-up, defined as clinical or image-based detection of tumour in treated breast or thoracic wall (local recurrence) or in the ipsilateral axilla or supraclavicular fossa or internal mammary chain (regional recurrence).
To compare the 5-years incidence of distant tumor recurrence between BA2 and BA3S | 5 years
  Distant recurrence rate occurring during the 5-years follow-up, defined as clinical or image-based detection of neoplastic affectation of other organs or tissues different from the treated breast, ipsilateral axilla or supraclavicular fossa or internal mammary chain.
To compare the acute and chronic toxicity of the two treatment modalities. | 5 years
  Toxicity, recorded using the Terminology Criteria for Adverse Events v4.0 (CTCAE).

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Algara Lopez, Medicine, Principal Investigator — Grupo de Investigación Clínica en Oncología Radioterápica (GICOR)
Locations (20):
- Spain (20):
  - Hospital Universitario de Araba, Vitoria-Gasteiz, Basque Country
  - Hospital Universitario de Cruces, Barakaldo, Bilbao
  - Hospital Universitario Sant Joan de Reus, Reus, Tarragona
  - Centro Oncológico de Galicia, A Coruña
  - Hospital Infanta Cristina, Badajoz
  - ICO Badalona, Badalona
  - Hospital Universitario Santa Lucía, Cartagena
  - Hospital Universitario de Donostia, Donostia / San Sebastian
  - ICO Girona, Girona
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario Gregrorio Marañón, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario Virgen de la Macarena, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital General Universitario de Valencia, Valencia

REFERENCES:
- [Background] Cortazar P, Zhang L, Untch M, Mehta K, Costantino JP, Wolmark N, Bonnefoi H, Cameron D, Gianni L, Valagussa P, Swain SM, Prowell T, Loibl S, Wickerham DL, Bogaerts J, Baselga J, Perou C, Blumenthal G, Blohmer J, Mamounas EP, Bergh J, Semiglazov V, Justice R, Eidtmann H, Paik S, Piccart M, Sridhara R, Fasching PA, Slaets L, Tang S, Gerber B, Geyer CE Jr, Pazdur R, Ditsch N, Rastogi P, Eiermann W, von Minckwitz G. Pathological complete response and long-term clinical benefit in breast cancer: the CTNeoBC pooled analysis. Lancet. 2014 Jul 12;384(9938):164-72. doi: 10.1016/S0140-6736(13)62422-8. Epub 2014 Feb 14. PMID 24529560
- [Background] Mamounas EP, Anderson SJ, Dignam JJ, Bear HD, Julian TB, Geyer CE Jr, Taghian A, Wickerham DL, Wolmark N. Predictors of locoregional recurrence after neoadjuvant chemotherapy: results from combined analysis of National Surgical Adjuvant Breast and Bowel Project B-18 and B-27. J Clin Oncol. 2012 Nov 10;30(32):3960-6. doi: 10.1200/JCO.2011.40.8369. Epub 2012 Oct 1. PMID 23032615
- [Background] Noh JM, Park W, Suh CO, Keum KC, Kim YB, Shin KH, Kim K, Chie EK, Ha SW, Kim SS, Ahn SD, Shin HS, Kim JH, Lee HS, Lee NK, Huh SJ, Choi DH. Is elective nodal irradiation beneficial in patients with pathologically negative lymph nodes after neoadjuvant chemotherapy and breast-conserving surgery for clinical stage II-III breast cancer? A multicentre retrospective study (KROG 12-05). Br J Cancer. 2014 Mar 18;110(6):1420-6. doi: 10.1038/bjc.2014.26. Epub 2014 Jan 30. PMID 24481403
- [Background] Shim SJ, Park W, Huh SJ, Choi DH, Shin KH, Lee NK, Suh CO, Keum KC, Kim YB, Ahn SD, Kim SS, Ha SW, Chie EK, Kim K, Shin HS, Kim JH, Lee HS. The role of postmastectomy radiation therapy after neoadjuvant chemotherapy in clinical stage II-III breast cancer patients with pN0: a multicenter, retrospective study (KROG 12-05). Int J Radiat Oncol Biol Phys. 2014 Jan 1;88(1):65-72. doi: 10.1016/j.ijrobp.2013.09.021. Epub 2013 Oct 22. PMID 24161425
- [Background] Nagar H, Boothe D, Ginter PS, Sison C, Vahdat L, Shin S, Smith M, Chao KS, Nori D, Hayes MK. Disease-free survival according to the use of postmastectomy radiation therapy after neoadjuvant chemotherapy. Clin Breast Cancer. 2015 Apr;15(2):128-34. doi: 10.1016/j.clbc.2014.09.012. Epub 2014 Nov 11. PMID 25459070
- [Background] Bernier J. Post-mastectomy radiotherapy after neodjuvant chemotherapy in breast cancer patients: A review. Crit Rev Oncol Hematol. 2015 Mar;93(3):180-9. doi: 10.1016/j.critrevonc.2014.10.011. Epub 2014 Oct 31. PMID 25465740
- [Background] White J, Mamounas E. Locoregional radiotherapy in patients with breast cancer responding to neoadjuvant chemotherapy: a paradigm for treatment individualization. J Clin Oncol. 2014 Feb 20;32(6):494-5. doi: 10.1200/JCO.2013.53.4974. Epub 2013 Dec 30. No abstract available. PMID 24378411
- [Background] Marks LB, Prosnitz LR. Reducing local therapy in patients responding to preoperative systemic therapy: are we outsmarting ourselves? J Clin Oncol. 2014 Feb 20;32(6):491-3. doi: 10.1200/JCO.2013.51.3523. Epub 2013 Dec 30. No abstract available. PMID 24378409
- [Background] Smith BD. Using chemotherapy response to personalize choices regarding locoregional therapy: a new era in breast cancer treatment? J Clin Oncol. 2012 Nov 10;30(32):3913-5. doi: 10.1200/JCO.2012.44.4539. Epub 2012 Oct 1. No abstract available. PMID 23032624
- [Background] Mamounas EP. Impact of neoadjuvant chemotherapy on locoregional surgical treatment of breast cancer. Ann Surg Oncol. 2015 May;22(5):1425-33. doi: 10.1245/s10434-015-4406-6. Epub 2015 Mar 2. PMID 25727558
- [Background] Rusthoven CG, Rabinovitch RA, Jones BL, Koshy M, Amini A, Yeh N, Jackson MW, Fisher CM. The impact of postmastectomy and regional nodal radiation after neoadjuvant chemotherapy for clinically lymph node-positive breast cancer: a National Cancer Database (NCDB) analysis. Ann Oncol. 2016 May;27(5):818-27. doi: 10.1093/annonc/mdw046. Epub 2016 Feb 9. PMID 26861597
- [Background] Belkacemi Y, Kaidar-Person O, Poortmans P, Ozsahin M, Valli MC, Russell N, Kunkler I, Hermans J, Kuten A, van Tienhoven G, Westenberg H; Breast Working Party of the EORTC Radiation Oncology Group (ROG). Patterns of practice of regional nodal irradiation in breast cancer: results of the European Organization for Research and Treatment of Cancer (EORTC) NOdal Radiotherapy (NORA) survey. Ann Oncol. 2015 Mar;26(3):529-35. doi: 10.1093/annonc/mdu561. Epub 2014 Dec 5. PMID 25480875
- [Background] Haffty BG, McCall LM, Ballman KV, McLaughlin S, Jagsi R, Ollila DW, Hunt KK, Buchholz TA, Boughey JC. Patterns of Local-Regional Management Following Neoadjuvant Chemotherapy in Breast Cancer: Results From ACOSOG Z1071 (Alliance). Int J Radiat Oncol Biol Phys. 2016 Mar 1;94(3):493-502. doi: 10.1016/j.ijrobp.2015.11.005. Epub 2015 Nov 10. PMID 26867878
- [Background] Arenas M, Montero A, de Las Penas MD, Algara M. The position and current status of radiation therapy after primary systemic therapy in breast cancer: a national survey-based expert consensus statement. Clin Transl Oncol. 2016 Jun;18(6):582-91. doi: 10.1007/s12094-015-1401-0. Epub 2015 Sep 14. PMID 26370420
- [Background] Dizon DS, Krilov L, Cohen E, Gangadhar T, Ganz PA, Hensing TA, Hunger S, Krishnamurthi SS, Lassman AB, Markham MJ, Mayer E, Neuss M, Pal SK, Richardson LC, Schilsky R, Schwartz GK, Spriggs DR, Villalona-Calero MA, Villani G, Masters G. Clinical Cancer Advances 2016: Annual Report on Progress Against Cancer From the American Society of Clinical Oncology. J Clin Oncol. 2016 Mar 20;34(9):987-1011. doi: 10.1200/JCO.2015.65.8427. Epub 2016 Feb 4. No abstract available. PMID 26846975
- [Background] Tsujimoto M, Nakabayashi K, Yoshidome K, Kaneko T, Iwase T, Akiyama F, Kato Y, Tsuda H, Ueda S, Sato K, Tamaki Y, Noguchi S, Kataoka TR, Nakajima H, Komoike Y, Inaji H, Tsugawa K, Suzuki K, Nakamura S, Daitoh M, Otomo Y, Matsuura N. One-step nucleic acid amplification for intraoperative detection of lymph node metastasis in breast cancer patients. Clin Cancer Res. 2007 Aug 15;13(16):4807-16. doi: 10.1158/1078-0432.CCR-06-2512. PMID 17699859
- [Background] Di Filippo F, Giannarelli D, Bouteille C, Bernet L, Cano R, Cunnick G, Sapino A. Elaboration of a nomogram to predict non sentinel node status in breast cancer patients with positive sentinel node, intra-operatively assessed with one step nucleic acid amplification method. J Exp Clin Cancer Res. 2015 Nov 4;34:136. doi: 10.1186/s13046-015-0246-2. PMID 26538019
- [Background] Navarro-Cecilia J, Duenas-Rodriguez B, Luque-Lopez C, Ramirez-Exposito MJ, Martinez-Ferrol J, Ruiz-Mateas A, Urena C, Carrera-Gonzalez MP, Mayas MD, Martinez-Martos JM. Intraoperative sentinel node biopsy by one-step nucleic acid amplification (OSNA) avoids axillary lymphadenectomy in women with breast cancer treated with neoadjuvant chemotherapy. Eur J Surg Oncol. 2013 Aug;39(8):873-9. doi: 10.1016/j.ejso.2013.05.002. Epub 2013 May 25. PMID 23711734
- [Background] Tamaki Y. One-step nucleic acid amplification assay (OSNA) for sentinel lymph node biopsy. Breast Cancer. 2015 May;22(3):230-4. doi: 10.1007/s12282-012-0390-x. Epub 2012 Aug 9. PMID 22875641
- [Background] Offersen BV, Boersma LJ, Kirkove C, Hol S, Aznar MC, Biete Sola A, Kirova YM, Pignol JP, Remouchamps V, Verhoeven K, Weltens C, Arenas M, Gabrys D, Kopek N, Krause M, Lundstedt D, Marinko T, Montero A, Yarnold J, Poortmans P. ESTRO consensus guideline on target volume delineation for elective radiation therapy of early stage breast cancer. Radiother Oncol. 2015 Jan;114(1):3-10. doi: 10.1016/j.radonc.2014.11.030. Epub 2015 Jan 24. PMID 25630428
- [Background] von Minckwitz G, Untch M, Blohmer JU, Costa SD, Eidtmann H, Fasching PA, Gerber B, Eiermann W, Hilfrich J, Huober J, Jackisch C, Kaufmann M, Konecny GE, Denkert C, Nekljudova V, Mehta K, Loibl S. Definition and impact of pathologic complete response on prognosis after neoadjuvant chemotherapy in various intrinsic breast cancer subtypes. J Clin Oncol. 2012 May 20;30(15):1796-804. doi: 10.1200/JCO.2011.38.8595. Epub 2012 Apr 16. PMID 22508812